CLINICAL TRIAL: NCT04097002
Title: A Phase I/IIa Study Evaluating the Safety and Tolerability of Intratumoral Administration of ORCA-010 in Treatment-Naïve Patients With Localized Prostate Cancer.
Brief Title: First in Man Clinical Study to Evaluate Safety and Tolerability of an Oncolytic Adenovirus in Prostate Cancer Patients.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Orca Therapeutics B.V. (Industry)
Collaborators: CMX Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CP-ORCA-010-02-CA; 2017-002737-39 (EudraCT Number); HC6-024-C227843 (Other: Health Canada)
Record Dates: First submitted 2019-08-02; First posted 2019-09-20 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Adenocarcinoma of the Prostate
Keywords: Prostate cancer; Intratumoral; ORCA; Adenovirus; Localized Prostate cancer; Intraprostatic
MeSH Terms: conditions — Prostatic Neoplasms; Adenoviridae Infections

STUDY DESIGN:
Intervention Model Description: Phase I and Phase IIa.
  Phase I/ Part A is a Single-escalated dose of ORCA-010 (3 dose cohorts) to determine the Maximum Tolerated Dose.
  Phase IIa/ Part B is a two administration dose cohort at Maximum Tolerated Dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase I, Part A, Cohort 1 (Experimental): Single dose-escalation of ORCA-010, Dose Cohort 1: 1x10*11 viral particles.
  Single dose of ORCA-010 will be administered for the first subject only and all relevant safety data for this subject will be reviewed by the DSMB prior to enrolling additional subjects.
  After the DSMB review, subjects will be enrolled in groups of three (including the first subject) and assessed for safety and Dose-Limiting Toxicity (DLT) after a single dose of ORCA-010.
  Group of 3 subjects.
  Dose will be escalated to the next cohort based on safety and toxicity results from the 3 treated subjects to determine the Maximum Tolerated Dose, if not determined by this cohort.
  Interventions: Biological: ORCA-010
- Phase I, Part A, Cohort 2 (Experimental): Single dose-escalation of ORCA-010, Dose Cohort 2: 5x10*11 viral particles.
  Group of 3 subjects.
  Dose will be escalated to the next cohort based on safety and toxicity results from the 3 treated subjects to determine the Maximum Tolerated Dose, if not determined by this cohort.
  Interventions: Biological: ORCA-010
- Phase I, Part A, Cohort 3 (Experimental): Single dose-escalation of ORCA-010, Dose Cohort 3: 1.5x10*12 viral particles.
  Group of 3 subjects.
  Dose will be considered as the Maximum Tolerated Dose based on safety and toxicity results from the 3 treated subjects.
  Interventions: Biological: ORCA-010
- Phase IIa, Part B, Cohort 4 (Experimental): Two dose administration of ORCA-010 seperated by 2 weeks, Dose Cohort 4: The Maximum Tolerated Dose depending on Phase I/ Part A results.
  Group of 12 subjects.
  Interventions: Biological: ORCA-010

INTERVENTIONS:
Biological: ORCA-010 — The investigational new drug ORCA-010 is a novel and improved oncolytic adenovirus based on the adenovirus serotype 5 (Ad5) genome. ORCA-010 replicates specifically in cancer cells and not in normal tissue cells. Its replication has been shown in a wide variety of cancer cell types, and it is not limited to prostate cancer.

SUMMARY:
This open label, dose escalating study is a phase I/IIa first in man study designed to evaluate the safety and tolerability of intratumoral administration of a novel oncolytic adenovirus (ORCA-010) in treating diagnosed treatment naïve Patients with localized prostate cancer.

DETAILED DESCRIPTION:
The study is divided into two parts. In Part A of the study, cohorts of subjects will be administered escalating doses of ORCA-010, using the 3+3 design. When the Maximum Tolerated Dose has been determined in Part A, a group of 12 new subjects will be treated in Part B of the study at this dose, with two administrations separated by a 2-week interval.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate, which is localized to the prostate ( within 24 months of screening)
2. Absence of lymph node, bone or other metastases as determined by MRI and CT scan, Bone Scan or nano-MRI (≤3 months prior to first administration)
3. Men between 18 and 75 years inclusive
4. ECOG status 0 or 1
5. Ability to understand and willingness to sign informed consent
6. Adequate liver, renal and bone marrow function: AST & ALT < 2.5 x ULN, total bilirubin < 1.5 x ULN, Alkaline phosphatase < 3 x ULN, Serum creatinine < 1.5 x ULN, Haemoglobin > 9.0 g/dL (5.59 mmol/L), Platelet count > 100x10*9/L, Neutrophils > 1.5x10*9/L, INR < 1.5xULN
7. eGFR ≥ 30 mL/min, using the Cockcroft - Gault Equation: Creatinine Clearance = [{(140 - age in years) x (weight in kg)} x 1.23] /serum Creatinine in Mmol/L

Exclusion Criteria:

1. Tumor not accessible for injection
2. Prior treatment of prostate cancer with radiation therapy or brachytherapy
3. Prior use of chemotherapy/hormone therapy for treatment of cancer
4. Target tumor adherent to a major vascular structure
5. Participation in any investigational drug study within the last 12 months prior to first administration of ORCA-010
6. Clinically significant active infection (viral or bacterial)
7. Known immunosuppressive diseases (e.g. HIV, Hepatitis B and C)
8. History of any other oncological malignancy, excluding basal cell carcinoma of the skin, in the past 5 years
9. Not willing to refrain from sexual activities or use a double barrier contraceptive device (condom with foam or vaginal suppository, diaphragm with spermicide) after administration of ORCA-010 and until 42 days after the last ORCA-010 administration
10. Severe obesity defined as Body Mass Index (BMI) > 30 kg/m2
11. Positive for adenovirus in throat swap or serum as determined by PCR at screening
12. Recent (within 3 months prior to enrolment in the study) history of alcohol abuse or other substances such as barbiturates, cannabinoids and amphetamines or a positive urine screen for drugs of abuse
13. Use of medication known to have immunosuppressive effects, except topical/inhaled steroids under 10 mg/day prednisolone equivalent (See Appendix 7)
14. Use of systemic antiviral medication within 3 months prior to enrolment in the study
15. Use of any anti-coagulants/blood thinner except for ASA 81mg
16. Any condition that in the opinion of the Investigator could interfere with the conduct of the study
17. For Part B only: Subjects enrolled in Part A of the study

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Treatment naïve men diagnosed with adenocarcinoma of the prostate,
Enrollment: 24 (Estimated)
Dates: Start 2019-11-12 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Safety profile of ORCA-010 | 365 days
  To evaluate safety and tolerability of intratumoral administration of ORCA-010 according to CTCAE V5.0. The primary endpoint of this study is to assess Dose Limiting Toxicities (DLTs) and the Maximum Tolerated Dose (MTD) for ORCA-010 to determine the final safety dose of administration for Phase IIa/Part B.

SECONDARY OUTCOMES:
Biological activity of ORCA-010 | 365 days
  To explore the biological activity of intratumoral administration of ORCA-010. Biological activity of ORCA-010 will be measured by assessing viral replication by measuring ORCA-010 virus DNA in blood. In addition, virus replication and spread will be assessed by staining prostate cancer tissue obtained through prostate biopsies with adenovirus specific antibodies. Subject's serum will be assayed for antibody responses against ORCA-010.
Antitumor immune responses | 365 days
  To evaluate potential antitumor immune responses following ORCA-010 administration. Subject's serum will be analyzed for antibody responses against tumor-associated antigens (e.g. PSA, PSMA, PCA3, and Prostein). Subject's Peripheral Blood Mononuclear Cells (PBMCs) will also be analyzed for cellular immune responses against tumor-associated antigens.
  Prostate biopsies will be taken to detect local antitumor immunological reactions (eg. infiltration and activation of T cells).
Shedding of ORCA-010 | 365 days
  Shedding of ORCA-010 will be assessed by detection of vector DNA in blood and urine using quantitative-PCR (Q-PCR).

CONTACTS AND LOCATIONS:
Overall Officials: Cornelis Groen, BSc Law, PhD, Study Director — Orca Therapeutics B.V.
Locations (5):
- Canada (5):
  - Jonathan Giddens Medicine Professional Corporation, Brampton, Ontario
  - G. Kenneth Jansz Medicine Professional Corporation, Burlington, Ontario
  - Research St. Joseph's - Hamilton, Hamilton, Ontario
  - The Fe/Male Health Centres Recruiting, Oakville, Ontario
  - Urology and Male Infertility Clinic, Scarborough Village, Ontario

IPD SHARING:
Plan to Share IPD: No
Not yet determined.